CLINICAL TRIAL: NCT05311462
Title: Exploration on Prevention and Treatment Mechanism of Obese Patient With Weight Cycling: An Investigator-initiated Single-center Cohort Study
Brief Title: An Observational Cohort Study to Obese Patients With Weight Cycling
Status: Active, not recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wei Chen, Professor, Peking Union Medical College Hospital
Other Study IDs: K3171
Record Dates: First submitted 2022-03-15; First posted 2022-04-05 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Weight Cycling; Obesity
MeSH Terms: conditions — Weight Cycling; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum samples, urine samples and fecal samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Weight-loss success with history of weight cycling: High-protein diet for three months
- Weight-loss failure with history of weight cycling: High-protein diet for three months

SUMMARY:
Medical nutritional weight loss was effective in reducing body weight and waist circumference and improving a range of cardiovascular disease risk factors in obese patients, with an average effective weight loss of 11.1 kg (about 13%) over 4 months in obese adults. However, it was found through the follow-up visit that these subjects had lost only 5.8kg from baseline and regained about half of their weight (5.1 kg, 48%) after 21 months of weight-loss intervention. In this study, intestinal flora analysis was proposed to identify the causes of individual repeated weight loss failure, structure changes of weight cycling and the advantage species of flora, and explore different intestinal microbiota（microbial genomics） in ending weight loss, obesity-related genetic characteristics (SNPs loci and RNA seq), metabolite（metabolomics）and potential interaction between appetite-related hormones and weight cycling triggers. This study aimed to provide new insights for implementing personalized weight loss programs to improve the success rate of weight loss. The obese patients who failed to lose weight repeatedly were recruited from Peking Union Medical College Hospital.

Research Contents:(1) Comparison of anthropometric, biochemical, energy consumption, and intestinal microbiota related indicators between groups; (2) Genotyping to screen out differential SNPs loci;(3) Analysis of the interaction between genes and environmental factors in different metabolic types of obesity. (4) A group of healthy volunteers with normal weight as the healthy control group.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight (18.5 ≤ BMI < 24 kg/m2) or obese (28 ≤ BMI < 35 kg/m2);
* Aged 18 to 50 years old;
* Han nationality;
* Able to follow the weight-loss prescription;
* Able to sign consent independently;
* Definition of Weight cycling: Loss weight more than once in the past 3 years, and weight regain exceeds 5% or more of the baseline weight of losing weight.

Exclusion Criteria:

* Bodyweight has changed more than ±10% in the past year;
* Taking drugs known to affect body weight (orlistat, GLP-1 receptor agonists, etc.);
* Taking drugs known to affect glucolipid metabolism (such as sulfonylureas, biguanides, acarbose, or insulin) have been taken in the past 6 months or at present; Lipid-lowering drugs such as statins, bate, niacin, and ezetimibe; Diuretics, β -blockers and other antihypertensive drugs; Glucocorticoid, thyroid hormone, etc.);
* Women who are currently pregnant or nearly 3 months breastfeeding;
* With serious eating disorders or vigorous exercise to lose weight;
* Hard physical workers;
* History of serious cardiovascular disease;
* Acute, chronic, or active gastrointestinal diseases;
* Serious systemic diseases;
* History of serious mental disorders;
* Cancer or active tumor;
* Secondary obesity or drug obesity patients: including hypothalamic obesity, pituitary obesity, hypercortisolism, and hypogonadism obesity;
* Severe liver dysfunction (ALT, AST, ALP, and TBil > the upper limit of 2.5 times reference value);
* Chronic kidney disease (eGFR < 60 mL/min/1.73 m2 or eGFR < 90 mL/min/1.73 m2 with proteinuria);
* Those who are considered by the researcher to be poor compliance or unable to complete this research well.

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Exposure group: Obese individuals with a history of weight cycling and successful weight loss with the nutritional intervention program after enrollment Control group: obese people with a history of previous weight cycle and failure to lose weight with nutritional intervention programs after enrollment Healthy control group: healthy volunteers of normal weight as a control population
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2025-01-20 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
BMI changes | Baseline time; after 1 months; after 45days; after 3 months; after 9 months；after1, 2, 3, 4 and 5 years
  Both the height and weight will be measured with a standard instrument and recorded in meters and kilograms respectively，following a requirement of accurating to two decimal places. And the weight and height will be combined to report in a form of BMI in kg/m^2.The changes in BMI before and after the study will be expressed as mean ± SD.
serum metabolome | Baseline time; after 9 months; after1, 2, 3, 4 and 5 years
  Collection of peripheral blood (PB) serum for metabolomics analysis PB will be collected directly into serum separation tubes. The serum samples from this study will be profiled by a non-targeted LC-MS based metabolomics analysis.Metabolomics will be profiled by reverse-phase LC-MS using C8-pos (reverse-phase C8 chromatography/positive and negative ion mode that detects non-polar and weak-polar compounds) and HILIC-pos (hydrophilic interaction chromatography/positive ion mode that detects polar molecules). This study will compare and observe the type and concentration difference of serum metabolites before and after.
Faecal metagenomes changes | Baseline time; after 45 days; after 3 months; after 9 months;after1, 2, 3, 4 and 5 years
  Patients will be requested to give stool samples that are collected in a sterile, sealed container and stored at -80 °C for strain-resolved metagenomic sequencing.DNA will be extracted from stool using the TIANamp Stool DNA Kit. We will conduct quality control using agarose gel electrophoresis. Metagenomics library will be constructed by NEXTflex Rapid DNA-Seq Kit (Illumina). The procedures included cluster generation, template hybridization, isothermal amplification, linearization, blocking and denaturation, and hybridization of the sequencing primers. We will observe differences in microbiome characteristics at various time points.
transcriptome changes | Baseline time; after 3 months;after1, 2, 3, 4 and 5 years
  Peripheral blood of the subjects will be collected and used to extract PBMC.RNA extraction and transcriptome sequencing of the PBMC samples will be used for transcriptome sequencing.Total RNA will be extracted by using the RNAeasy kit according to the manufacturer's instructions. The purity, concentration, and integrity of total RNA will be checked using the NanoPhotometer spectrophotometer, the Qubit RNA Assay Kit in Qubit 2.0 Fluorometer and the RNA Nano 6000 Assay Kit of the Bioanalyzer 2100 System, respectively. Besides, RNA degradation and contamination will be monitored on 1% agarose gels. Sequencing libraries will be generated using the rRNA-depleted RNA by NEBNext UltraTM Directional RNA Library Prep Kit for Illumina and sequenced on an Illumina HiSeq 4000 platform. Transcriptome changes before and after the intervention will be observed to predict the outcome of weight-loss interventions.

OTHER OUTCOMES:
insulin resistance index | Baseline time; after 3 months; after 9 months;after1, 2, 3, 4 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chen, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li W, Wang D, Chen H, Liu Y, Dong S, Sun M, Chen W. The relationship between psychological distress and weight maintenance in weight cycling: mediating role of eating behavior. BMC Public Health. 2024 Mar 26;24(1):894. doi: 10.1186/s12889-024-18349-5. PMID 38532390